CLINICAL TRIAL: NCT01877928
Title: Use of the Boussignac CPAP System Immediately Following Extubation to Improve Lung Function in Adults With Moderate to Severe Obstructive Sleep Apnea
Brief Title: Post-extubation Boussignac CPAP System in Adults With Moderate to Severe Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Most OSA patients were not obese and/or admitted over night so the study was not feasible.
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Kim Turner, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMED-079-12; 6006956 (Other: Institutional Research Ethics board database)
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Obstructive sleep apnea, CPAP, Boussignac
MeSH Terms: conditions — Sleep Apnea, Obstructive; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Boussignac CPAP device (Experimental): Patients previously diagnosed with obstructive sleep apnea and who are undergoing abdominal or peripheral surgery will have the Boussignac CPAP mask applied for 1 hour starting immediately post-extubation
  Interventions: Device: Boussignac CPAP device
- standard CPAP (Active Comparator): Patients previously diagnosed with obstructive sleep apnea who are undergoing peripheral or abdominal surgical procedures will receive the standard-of-care for obstructive sleep apnea. This typically involves CPAP application only at night
  Interventions: Device: standard CPAP

INTERVENTIONS:
Device: Boussignac CPAP device — Is a continuous positive airway pressure (CPAP) system marketed in Canada and the US for the treatment of Obstructive Sleep Apnea. The main difference is that this system is portable wheres the standard hospital CPAP is not. This allows for the application immediately post-extubation.
  Other Names: Boussignac CPAP device,
  Arms: Boussignac CPAP device
Device: standard CPAP — Standard of care postoperative treatment for OSA.
  Other Names: standard of care CPAP
  Arms: standard CPAP

SUMMARY:
The purpose of this study is to assess the efficacy of the Boussignac positive airway pressure system (a mask) applied immediately following post-operative extubation in improving lung function in patients with obstructive sleep apnea (OSA). Assessments will be done before surgery and then at 1, 2 and 24 hours following extubation and will be compared to standard care for perioperative airway support. The study aims to give a broader and more inclusive picture (than the current literature) in terms of whether the Boussignac CPAP system should be considered for utilization by anesthesiologists caring for surgical patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

-> 18 years of age

* ASA II-IV
* Previous diagnosis of moderate to severe obstructive sleep apnea
* diagnosed via polysomnography
* BMI < 40
* scheduled for an abdominal or peripheral surgical procedure requiring endotracheal intubation and admission to hospital

Exclusion Criteria:

* BMI > 40
* Age <18 years
* inability to provide signed informed consent
* intra-thoracic
* head or neck surgery
* contraindication for immediate post-extubation application of CPAP
* not expected to be eligible for timely extubation following the surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
percent forced vital capacity %(FVC) | 24 hours postoperatively
  %FVC will be assessed 24 hours postoperatively in patients who received the Boussignac CPAP mask immediately post-extubation and these values compared to those of patients who received the standard-of-care treatment for obstructive sleep apnea

SECONDARY OUTCOMES:
% forced expiratory volume in 1 second (FEV1) | 1,2 and 24 hours post-operatively

OTHER OUTCOMES:
Peak expiratory flow rate (PEFV) | 1,2 and 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kim E Turner, MD, FRCPC, Principal Investigator — Queen's University & Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada